CLINICAL TRIAL: NCT04099290
Title: Circulating Tumor DNA (ctDNA) in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: American Society of Clinical Oncology (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 1835; 5K12CA120780-15 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Neoplasm; Carcinoma, Squamous Cell
Keywords: Squamous Cell Carcinoma; Circulating Tumor DNA
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and tumor samples — Blood samples to be obtained at consent, post-operatively, post-adjuvant treatment, and at follow-up or recurrence. Tumor samples to be obtained at surgery and at time of recurrence or post-treatment biopsy, if applicable.

SUMMARY:
Circulating tumor DNA (ctDNA) is a blood-based test that measures dying or dead cancer cells that are already circulating in the blood. In this study, the investigators will enroll patients who are planning to receive surgery to remove their head and neck cancer. The investigators are interested to learn how ctDNA levels change with surgery and over the course of time. The investigators also want to determine if there are certain features of the tumor or the patient themselves that might cause ctDNA to be higher than other patients. Also, the investigators want to explore if the detection of ctDNA following surgery is related to cancer recurrence.

DETAILED DESCRIPTION:
The investigators will take a piece of the tumor from the surgery and determine if they can identify mutations, or changes in the genetic makeup of the cells due to cancer, that are specific to the tumor. Based on this information, the investigators will design a test using PCR, which is a technology that allows for the amplification of the DNA, that is specific to the mutation identified in the tumor. Once verified, the presence (or absence) of ctDNA in the blood can be measured. The investigators will measure this blood test prior to surgery and at multiple time points following surgery. Specimens will be collected at the time of planned clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information. Consent for the use of any residual material from biopsy and/or surgical resection (archival tissue) and serial blood draws will be required for enrollment.
* Age ≥ 18 years of age on day of signing informed consent
* Newly diagnosed, histologically confirmed squamous cell carcinoma of the head and neck, including the following subtypes: oral cavity, oropharynx, larynx
* Must be planning to undergo gross total resection of the primary tumor with curative intent at UNC-CH hospital
* No prior, definitive therapy to primary tumor. Must meet one of the following clinical stages: T3-T4 (if T1/T2 must have nodal involvement), Any N, M0
* Patient must be amenable to receiving adjuvant therapy with radiotherapy +/- systemic therapy, as clinically indicated, based on either standard of care (SOC) or appropriate clinical trial.
* Diagnostic tumor material must be available for correlative analysis
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee

Exclusion Criteria:

* Has known evidence of metastatic disease based on clinical or radiographic studies
* Women who are pregnant or nursing
* History of another primary malignancy in the last 5 years prior to registration. Patients with history of in situ cancer or basal or localized squamous cell skin cancers are eligible.
* Patients with primary skin cancers of the head and neck, including basal or squamous cell cancers
* Prior chemotherapy, IP, biologic, or hormonal therapy for HNSCC treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Head and Neck Cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of tumor-specific mutation in pre-operative circulating tumor DNA of patients with locally-advanced HNSCC who are receiving surgery for treatment of their primary tumor | Time of consent

SECONDARY OUTCOMES:
Rate of tumor-specific mutation in post-operative circulating tumor DNA in patients with locally-advanced HNSCC who received surgery for treatment of their primary tumor | Post-surgery/pre-treatment, post-surgery/post-treatment (approximately 6 weeks following initiation of treatment and every 3 months up to 2 years), and at disease recurrence if applicable (up to 5 years)
Change in ctDNA levels (i.e., copies per mL plasma) over time | Time of consent, post-operatively (approximately 1-4 weeks after surgery), post-adjuvant treatment (approximately 6 weeks following initiation of treatment) and follow-up (every 3 months up to 2 years)/recurrence if applicable (up to 5 years)
Description of tumor-specific mutations in surgical specimens by NGS | Surgery and post-treatment biopsy/recurrence if applicable(up to 5 years)
Correlation between post-operative plasma ctDNA levels and surgical margins | Post-operatively (approximately 1-4 weeks after surgery)
Correlation between post-operative plasma ctDNA levels and extra-capsular extension | Post-operatively (approximately 1-4 weeks after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, MD, Principal Investigator — UNC Health Care; Gaorav Gupta, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States